CLINICAL TRIAL: NCT00003907
Title: Chemoembolization in Hepatocellular Carcinoma or Neuroendocrine Hepatic Metastases: A Phase II Multi-Center Trial
Brief Title: Chemoembolization in Treating Patients With Primary Liver Cancer or Metastases to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067083; U10CA021115 (NIH); E4298 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 1999-11-01; First posted 2003-10-09 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma; liver metastases
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Cisplatin; Platinum; Doxorubicin; Mitomycin; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepatocellular carcinoma (Experimental): Chemoemulsion (doxorubicin, mitomycin and cisplatin) followed by embolization. The entire procedure will be repeated separately to each involved lobe beginning within 8 weeks of the last lobar chemoembolization.
  Interventions: Drug: cisplatin; Drug: doxorubicin; Drug: mitomycin; Procedure: embolization
- Neuroendocrine hepatic metastases (Experimental): Chemoemulsion (doxorubicin, mitomycin and cisplatin) followed by embolization. The entire procedure will be repeated separately to each involved lobe beginning within 8 weeks of the last lobar chemoembolization.
  Interventions: Drug: cisplatin; Drug: doxorubicin; Drug: mitomycin; Procedure: embolization

INTERVENTIONS:
Drug: cisplatin — Doxorubicin 30 mg, mitomycin 30 mg, and cisplatin 100 mg (all in powdered form) should be dissolved in 10-15 cc of contrast agent (such as isovue or optiray).
  Other Names: Cis-diaminedichloroplatinum Cis-diaminedichloroplatinum (II),; diaminedichloroplatinum,; cis-platinum,; platinum,; Platinol,; Platinol-AQ,; DDP,; CDDP,; DACP,; NSC 119875
Drug: doxorubicin — Doxorubicin 30 mg, mitomycin 30 mg, and cisplatin 100 mg (all in powdered form) should be dissolved in 10-15 cc of contrast agent (such as isovue or optiray).
  Other Names: Adriamycin,; Rubex,; Adriamycin RDF,; Adriamycin PFS,; hydroxydaunorubicin,; hydroxydaunomycin,; ADR
Drug: mitomycin — Doxorubicin 30 mg, mitomycin 30 mg, and cisplatin 100 mg (all in powdered form) should be dissolved in 10-15 cc of contrast agent (such as isovue or optiray).
  Other Names: Mutamycin,
Procedure: embolization — Immediately following delivery of the chemoemulsion, particulate embolization is performed. The particulate embolic material is prepared on a separate table or tray, using absorbable gelatin sponge (Gelfoam, Upjohn, Kalamazoo, MI), in either powder or pledget form. Approximately 1 g of this temporary occlusive agent is dissolved in 20-30 cc of full-strength contrast with 2.4 cc of absolute alcohol.
  Other Names: trans-arterial chemoembolization,; TACE

SUMMARY:
RATIONALE: Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor.

PURPOSE: Phase II trial to study the effectiveness of chemoembolization in treating patients who have primary liver cancer or metastases to the liver that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate time to progression of disease in patients with unresectable hepatocellular carcinoma or neuroendocrine hepatic metastases undergoing chemoembolization.
* Evaluate tumor response achievable with chemoembolization in this patient population.
* Evaluate the toxicities of this treatment in these patients.
* Evaluate survival of these patients following this treatment.
* Evaluate extrahepatic patterns of failure following chemoembolization, to determine whether intrahepatic progression may be forestalled and survival affected in these patients.
* Validate a consistent method of performing chemoembolization in a multicenter setting.

OUTLINE: Patients are stratified according to disease (hepatocellular carcinoma vs neuroendocrine hepatic metastases).

Patients undergo placement of a visceral arterial catheter. Patients receive doxorubicin, mitomycin, and cisplatin as a chemoemulsion via the arterial catheter into 1 hepatic lobe only. Immediately following delivery of the chemoemulsion, particulate embolization is performed. The opposite lobe, if involved, is treated within 3-5 weeks of treatment of the initial lobe.

In the absence of unacceptable toxicity, each involved lobe is treated separately a second time, in the same sequence, beginning 8 weeks after the last lobular chemoembolization. After completion of all protocol therapy, retreatment on study of either lobe is allowed for regrowth, recurrence, or new disease, provided at least 3 months have elapsed since the initial treatment of that lobe.

Patients are followed for 5 years.

PROJECTED ACCRUAL: A total of 19-42 patients will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven intrahepatic hepatocellular carcinoma or neuroendocrine tumor.
* Unresectable.
* Bidimensionally measurable disease by Computed Tomography (CT), Magnetic resonance imaging (MRI), or UltraSound Scanning (US) within 6 weeks of registration.
* Evidence of patent portal vasculature by Doppler US, MRI, or angiography.
* Serum total bilirubin < 2.0 mg/dl and serum creatinine < 2.0 mg/dl within 4 weeks of registration.
* Absolute neutrophil count (ANC) > 2000/µl and platelets > 50,000/µl within 4 weeks of registration.
* Expected survival of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Age >= 18 years.

Exclusion Criteria:

* Evidence of extrahepatic disease that is likely to be life-threatening within 3 months, such as brain or symptomatic lung metastases.
* Previous intra-arterial or intra-hepatic chemotherapy or prior systemic chemotherapy within 4 weeks.
* Concurrent malignancy.
* Pregnant or breast-feeding women.
* History of life-threatening contrast allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1999-12-15 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith E. Stuart, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (37):
- United States (37):
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG membership institution between August 6, 1999 and September 15, 2006. The first patient was accrued on December 15, 1999.
Period: Overall Study
Arm/Group | Hepatocellular Carcinoma | Neuroendocrine Hepatic Metastases
Started | 19 | 31
Eligible | 18 | 29
Received Protocol Therapy (Treated) | 18 | 31
Eligible and Treated | 17 | 29
Completed | 6 | 8
Not Completed | 13 | 23
Not completed — Adverse Event | 2 | 11
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Progressive disease | 4 | 4
Not completed — Complicating disease | 1 | 0
Not completed — Other | 1 | 3
Not completed — ineligible or not treated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hepatocellular Carcinoma | Neuroendocrine Hepatic Metastases | Total
Number analyzed (Participants) | 17 | 29 | 46
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 81] | 62 [28 to 83] | 62 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 15 | 19
  Male | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  United States | 17 | 29 | 46

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression was defined as time from embolization to documented disease progression. Patients without documented progression were censored at the time of the last documented disease evaluation or of the last treatment ended, whichever was more recent.Disease progression was defined as significant increase in size of lesions or appearance of new metastatic lesions. Specifically, 1) >=25% increase in the area of any malignant lesions greater than 2 cm² or in the sum of the products of the individual lesions in a given organ site; 2)>=50% increase in the size of the product of diameters if only one lesion is available for measurement and was less than or equal to 2 cm² in size at the initiation of therapy; 3)>=25% increase in the sum of the liver measurements below the costal margins and xyphoid; 4)Appearance of new malignant lesions
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 year.
Population: All eligible and treated patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Hepatocellular Carcinoma | Neuroendocrine Hepatic Metastases
Number analyzed (Participants) | 17 | 29
Months | 2.3 [1.1 to 24.0] | 7.2 [4.4 to 17.3]

2. Secondary Outcome: Tumor Response
Description: Clinical complete response was defined as complete disappearance of all clinically detectable malignant disease for at least 4 weeks. Partial response was defined as >= 50% decrease in tumor size for at least 4 weeks without increase in size of any area of known malignant disease of greater than 25%, or appearance of new areas of malignant disease. Tumor response was defined as complete response + partial response.
Time Frame: Assessed every 6 weeks
Population: all eligible and treated patients
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Hepatocellular Carcinoma | Neuroendocrine Hepatic Metastases
Number analyzed (Participants) | 17 | 29
Proportion of participants | 0 [0 to 0.16] | 0.17 [0.07 to 0.33]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from registration to death from any causes.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 year.
Population: all eligible and treated patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Hepatocellular Carcinoma | Neuroendocrine Hepatic Metastases
Number analyzed (Participants) | 17 | 29
Months | 12.0 [3.9 to 27.6] | 21.2 [9.7 to 38.1]

ADVERSE EVENTS:
Time Frame: Assessed every cycle (each chemo-embolization procedure is considered a cycle) while on treatment and for 30 days after the end of treatment.
Arm/Group | Hepatocellular Carcinoma | Neuroendocrine Hepatic Metastases
Serious Adverse Events (participants affected / at risk) | 18/18 | 30/31
Other Adverse Events (participants affected / at risk) | 18/18 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hepatocellular Carcinoma (N=18) | Neuroendocrine Hepatic Metastases (N=31)
Anemia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Neutrophils, decreased) (Investigations) | 1 | 2
Thrombocytopenia (Platelets, decreased) (Investigations) | 2 | 0
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular arrhythmias (Cardiac disorders) | 0 | 1
Acute vascular leak syndrome (Vascular disorders) | 0 | 1
Cardiac-ischemia (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 2 | 4
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 1
Operative injury of vein/artery (Injury, poisoning and procedural complications) | 0 | 2
Fever (General disorders) | 1 | 0
Weight gain (Investigations) | 2 | 0
PT (Investigations) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 7
Vomiting (Gastrointestinal disorders) | 0 | 1
Hemorrhage with grade 3 or 4 platelets (Vascular disorders) | 1 | 0
GI-other (Gastrointestinal disorders) | 0 | 1
Melena/GI bleeding (Gastrointestinal disorders) | 1 | 1
Alkaline phosphatase (Investigations) | 1 | 3
Bilirubin (Investigations) | 4 | 1
Hepatic enlargement (Hepatobiliary disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 4
Liver dysfunction/failure (Hepatobiliary disorders) | 2 | 2
SGOT (Investigations) | 18 | 26
SGPT (Investigations) | 0 | 6
Hepatic-other (Hepatobiliary disorders) | 0 | 3
Infection w/o neutropenia (Infections and infestations) | 1 | 1
Hypercholesterolemia (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Arachnoiditis (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Dizziness/lightheadedness (Nervous system disorders) | 0 | 1
Infection-other (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatinine (Investigations) | 1 | 2
Renal failure (Renal and urinary disorders) | 2 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hepatocellular Carcinoma (N=18) | Neuroendocrine Hepatic Metastases (N=31)
Anemia (Blood and lymphatic system disorders) | 16 | 21
Leukopenia (Leukocytes, decreased) (Investigations) | 3 | 7
Neutropenia (Neutrophils, decreased) (Investigations) | 0 | 6
Thrombocytopenia (Platelets, decreased) (Investigations) | 11 | 14
Edema (Skin and subcutaneous tissue disorders) | 2 | 1
Fatigue (General disorders) | 9 | 16
Fever (General disorders) | 7 | 9
Rigors/chills (General disorders) | 1 | 3
Weight loss (Investigations) | 3 | 11
PT (Investigations) | 10 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 13
Ascites (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 10 | 21
Vomiting (Gastrointestinal disorders) | 7 | 21
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 8
Alkaline phosphatase (Investigations) | 15 | 24
Bilirubin (Investigations) | 7 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 | 17
Abdominal pain (Gastrointestinal disorders) | 1 | 13
Hepatic pain (Hepatobiliary disorders) | 2 | 1
Pain-other (General disorders) | 3 | 1
Creatinine (Investigations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No